CLINICAL TRIAL: NCT03136211
Title: A Hybrid Effectiveness-Implementation Trial of a Complex Multiple Risk Intervention to Promote Healthy Behaviors in People Between 45 to 75 Years Attended in Primary Health Care
Brief Title: Complex Multiple Risk Behavior Intervention in People Between 45 to 75 Years (EIRA Study)
Acronym: EIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Department of Health, Generalitat de Catalunya (Other Government); Parc Sanitari Sant Joan de Déu (Other); Sanidad de Castilla y León (Other); Servei de Salut de les Illes Balears (Unknown); Institut Català de la Salut (Other); Servicio Aragones De Salud (Other); Osakidetza (Other); Andaluz Health Service (Other Government); Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other); Servicio Gallego de Salud (Other Government)
Responsible Party: Principal Investigator, Bonaventura Bolíbar Ribas, redIAPP Coordinator, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4R15/032; PI15/00114 (Other Grant/Funding Number: Instituto de Salud Carlos III. Ministry of Economy, Industry and Competitiveness); SLT002/16/00112 (Other Grant/Funding Number: Department of Health of the Government of Catalonia.)
Record Dates: First submitted 2017-04-07; First posted 2017-05-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Health Behavior; Health Promotion; Primary Health Care; Implementation Research; Smoking Cessation; Mediterranean Diet; Physical Activity
MeSH Terms: conditions — Health Behavior; Smoking Cessation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EIRA intervention (Experimental): EIRA intervention It is based on the Transtheoretical Model (TTM) and States of Change and it is made by physicians and nurses in routine care of primary care practices according to the conceptual framework of the "5A": Ask, Advise, Assess, Assist, and Arrange. It consists of a first visit of screening ("Ask"). Subsequently, the professional develops a personalized plan that is negotiated with the participant ("Advise" and "Assess"). This plan is reviewed during successive visits and positive changes are reinforced and new objectives are negotiated ("Assist" and "Arrange"). The motivational interview is the essential tool of the intervention. The intervention is carried out to different levels: individual, group and community.
  Interventions: Behavioral: EIRA intervention
- Usual care (No Intervention): Health providers of this group integrate in their practice the recommendations of the Program of Preventive Activities and Health Promotion (PAPPS)". These guidelines are based on systematic screening and brief advice for the prevention of cardiovascular and mental diseases and cancer as well as vaccine recommendations.

INTERVENTIONS:
Behavioral: EIRA intervention — Individual intervention has an average intensity between 2 and 3 visits; if necessary, professionals have the freedom to make a greater number of visits. Group intervention is carried out through health education workshops. These workshops take place 15-20 days after initiating the individual intervention and they are conducted by primary care providers in the health center. A group of 12-15 people attend in each workshop. Community intervention focuses mainly on the social prescription of resources and activities that are carried out in the community where the participant person resides. In addition the intervention has the support of information and communication technologies, such as a web addressed to the participant, a mobile app or the sending personalized text messages.
  Arms: EIRA intervention

SUMMARY:
This study examines the effectiveness and the costs of a complex multiple risk behavior intervention to promote healthy behaviors in people aged between 45 and 75 years attended in Primary Health Care services. This intervention aims to reduce tobacco use, to enhance adherence to the Mediterranean dietary pattern and to increase physical activity. The study also seeks to provide evidence on the strategies to integrate health promotion into the usual clinical practice of primary care providers.

DETAILED DESCRIPTION:
Health promotion interventions are complex and need in-depth understanding of the context which is part of its effect. In this respect, the methodology proposed by the Medical Research Council offers a unique opportunity. This methodology proposes a development in five sequential phases in which both quantitative and qualitative methods are used, which include: a) definition of the theoretical basis (preclinical phase), b) modeling (phase I), c) exploratory trial (phase II), d) definitive randomized controlled trial (phase III) and e) long-term implementation (phase IV). This methodology promotes the participation of citizens and professionals in research and increases the acceptability and the feasibility of intervention. It is also an ideal tool to achieve the sustainability of interventions and the transfer of research to practice. Research on complex interventions marks a turning point in the conventional way of conducting experimental studies in which the most important thing is finding value and understanding the context of practice rather than trying to control its influence. Hybrid trials represent the ideal design because they allow a joint assessment of clinical effectiveness and implementation, thanks to their dual approach.

In this connection, the researchers started in 2012 the EIRA study and carried out the first three phases (preclinical phase, phase I and phase II). Currently, researchers are pursuing the phase III whose purpose is to assess the cost-effectiveness and the implementation of a health promotion intervention through a hybrid design.

This cluster randomized controlled trial aims to assess the effectiveness and the implementation of a complex multiple risk behavior intervention with two parallel groups (intervention and usual care). It is based on:

* The "Consolidated Framework for Implementation Research" (CFIR) which identifies five constructs: 1) intervention characteristics (intervention source, evidence strength and quality, relative advantage, adaptability, trialability, complexity, design quality and packaging; and cost); 2) outer setting (patient needs and resources, cosmopolitanism, peer pressure, and external policy and incentives); 3) inner setting (structural characteristics, networks and communications, culture, implementation climate and readiness for implementation); 4) characteristics of individuals (knowledge and beliefs about the intervention, self-efficacy, individual state of change, individual identification with the organization, and other personal attributes); and 5) the implementation process itself.
* A set of discrete implementation strategies which includes: plan strategies (gather information, adapt and pilot material and processes, build buy-in, initiate leadership and develop relationships); educate strategies (develop materials, educate, educate through peers, inform and influence stakeholders); finance strategies (modify incentives and facilitate financial support); restructure strategies (revise professional roles and create community and group interventions committees) and quality management strategies (develop and organize implementation monitoring systems, conduct continuous assessment and feedback, establish a system of reminders, obtain and use patient opinion, centralize technical assistance focused on implementation issues).
* An evaluation framework to determine the success of implementation.

The study will be carried out in three stages:

STAGE 1: PRE-IMPLEMENTATION. During this stage, the researchers will assess local needs and resources to develop specific implementation strategies. Likewise, the scientific literature will be reviewed and the perspectives of clinicians on the internal resources will be measured by the "Survey of Organizational Attributes for Primary Care". All the support material for the intervention will be drawn up, besides the facilitator (member of the research team) and the leader (member of the primary care team) of the implementation will be designated. Mechanisms for the effective communication and the case report form (CRF) will be defined and piloted. Formal compromises will be made with the managers (at the macro, meso and micro levels) and with the professionals involved. Training activities will be carried out in which training in motivational interview will have a central role. In addition, a checklist (on-line database) will be developed and piloted to monitor the progress of implementation in each primary care center.

STAGE 2: IMPLEMENTATION. In this stage the implementation plan will be carried out. The facilitator and the leader of implementation will monitor the implementation processes, identify opportunities for improvement and optimize implementation. Likewise, positive feedback techniques will be used towards the main stakeholders in order to keep the agreed compromise and the motivation. Besides, health professionals will receive continuous training in motivational interview.

STAGE 3: POST-IMPLEMENTATION.

The evaluation of the implementation will be carried out through qualitative and quantitative research. It will be evaluated in terms of:

A) OUTCOMES (see section "Outcome Measures"). B) DETERMINANTS. Three focus groups (one of health professionals and two of participants) will be conducted in each health center. Sampling will be theoretical (discursive plurality). Sessions will be transcribed in an anonymous fashion. A thematic content analysis will be done. The CFIR constructs will be scored following standard criteria that they will reflect the influence of the construct on the implementation (positive or negative) and its magnitude (between 1 and 2).

C) LEVEL OF DEVELOPMENT. The level of development of each of the implementation strategies will be determined from the online database. Updating of this database will be carried out by the facilitator of implementation. Likewise, logistic regression models will be developed in which the dependent variable will be the effectiveness of the intervention, considered as a positive change in any of the three behaviors studied. In one of the models the independent variables will be the quantitative measures of the results of the implementation and in the other, the degree of implementation of the different strategies. The purpose of these analyzes is to model the relationship between the implementation variables and those of effectiveness. On the other hand, the influence and the magnitude of the determinants of the implementation and the results will be established through multivariate models.

SAMPLE SIZE It will be necessary to study a minimum of 3640 people (1820 for each of the two groups). This sample size will allow to detect an increase of 8% in the proportion of people who show a positive change in one or more of the three behaviors in the intervention group over control group. The proportion of losses during follow-up estimated was of 30%. The sample size was decided taking into account the effect of design (intraclass correlation coefficient of 0.01).The power was 80% and alpha risk 5%.

ELIGIBILITY:
Inclusion Criteria:

* People who carry out 2 or more of the following unhealthy behaviors: tobacco consumption, low adherence to the Mediterranean dietary pattern or insufficient physical activity. In addition, they must have a professional provider of the health center assigned and voluntarily agree to participate.

Exclusion Criteria:

* Advanced serious illnesses
* Cognitive impairment
* Dependence in basic everyday activities
* Severe mental illness
* People included in a long term home health care program
* People in treatment for cancer
* People in end-of-life care

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3062 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Positive change in baseline eating behavior | at the study entry and at 12 months
  Adherence to the Mediterranean dietary pattern in low adherence people. For the evaluation, the 14-item Questionnaire of Mediterranean diet adherence (PREDIMED study) will be used.
Effectiveness: Positive change in baseline physical activity behavior | at the study entry and at 12 months
  Sufficient physical activity in insufficiently active people. For the evaluation, the "International Physical Questionnaire (IPAQ)" will be used.
Effectiveness: Positive change in baseline smoking behavior | at the study entry and at 12 months
  Smoking cessation in smokers. For the evaluation, the interview will be used and the cooximetry (optional).
Implementation: adoption | Within 2 months prior to the start of the intervention
  Proportion of professionals who express their willingness to participate in the study between of total of potential professionals.
Implementation: early acceptability | Within 2 months prior to the start of the intervention
  They will be evaluated in professionals and participants by means of a survey.
Implementation: final acceptability | at 12 months post intervention
  They will be evaluated in professionals and participants by means of a survey. What is more, discussion groups will be held at the end of the intervention with the professionals and participants.
Implementation: early appropriateness | Within 2 months prior to the start of the intervention
  They will be evaluated in professionals and participants by means of a survey.
Implementation: final appropriateness | at 12 months post intervention
  They will be evaluated in professionals and participants by means of a survey. What is more, discussion groups will be held at the end of the intervention with the professionals and participants.
Implementation: Cost of time invested in training and organizational meetings | at 12 months post intervention
  Cost of time invested in training and organizational meetings to carry out the intervention.
Implementation: feasibility | at 12 months post intervention
  On the basis of the calculation of participation, recruitment and retention rate.
Implementation: fidelity of the motivational interview technique | Within 2 months prior to the start of the intervention
  The quality of the motivational interview will be evaluated through videotapes of visits to simulated patients through the "motivational interviewing assessment scale".
Implementation: fidelity of the planned intervention | at 12 months post intervention
  The degree of compliance of the activities recorded in the case report form will be analyzed.
Implementation: penetration | Within six months of the end of intervention
  The proportion of professionals who have integrated the intervention into their usual clinical practice within six months of the end of intervention.

SECONDARY OUTCOMES:
Effectiveness: Beginning or making of a behavior change | at the study entry and at 12 months
  Proportion of people who are in the stages of action, maintenance or termination according to the transtheoretical model at the entry and at the end of the study.
Effectiveness: Change from baseline on arterial stiffness at 12 months | at the study entry and at 12 months.
  Arterial stiffness assessed by the "Cardio-Ankle Vascular Index (CAVI)". CAVI will be measured in the routine clinical practice by the Vascular Screening System VaSera VS-1500N.
Change from baseline on health-related quality of life | at the study entry and at 12 months.
  Health-related quality of life as measured by the EuroQol-5D questionnaire.
Change from baseline on costs of number visits, diagnostic tests, community resources used and loss of productivity | at the study entry and at 12 months.
  Number in the last 12 monts of: primary-care and specialists visits, outpatient diagnostic tests, community resources used, group sessions attended and days off work per participant

OTHER OUTCOMES:
Effectiveness: Reduction of the cardiovascular risk | at the study entry and at 12 months
  Proportion of people with low/moderate and high/very high baseline cardiovascular risk who have reduced it by 10% and 25% respectively. Cardiovascular risk will be calculated using REGICOR and SCORE function charts.
Effectiveness: Reduction of the risk of depression | at the study entry and at 12 months
  Effect size greater than or equal to 8% in the probability of risk of depression in people with moderate to high risk of depression at the entry of study. People have received usual care will be compared to those who received the EIRA intervention. Risk of depression will be calculated using the algorithm PredictD.
Effectiveness:change from baseline on body mass index | at the study entry and at 12 months.
  Body mass index is defined as the body weight divided by the square of the body height, and is expressed in units of kg/m2.
Effectiveness:change from baseline on waist circumference | at the study entry and at 12 months.
  The waist circumference will be measured at a level midway between the lowest rib and the iliac crest. It will be expressed in units of cm.
Effectiveness:change from baseline on blood pressure | at the study entry and at 12 months.
  It will be measured in the routine clinical practice by validated electronic monitors and it will be expressed in units of mmHg.
Effectiveness:change from baseline on lipid profile | at the study entry and at 12 months.
  The lipid profile will include: low-density lipoprotein (LDL), high-density lipoprotein (HDL), triglycerides and total cholesterol. They will be expressed in units of mg/dl.
Effectiveness: change from baseline on ankle-brachial index | at the study entry and at 12 months.
  It will be measured in the routine clinical practice by the Vascular Screening System VaSera VS-1500N.
Effectiveness: change from baseline on the "REgicor and Artper Score fOr aNkle brachial index (REASON)" | at the study entry and at 12 months.
  REASON is a validated screening test to select candidates for ankle-brachial index (ABI) measurement in the Spanish population. It uses clinical data routinely collected in general practice for cardiovascular risk estimation. This test integrates the following measures: personal history of hypercholesterolemia, diabetes mellitus, arterial hypertension, smoking, body mass index, blood pressure, glycaemia, total cholesterol, high density lipoprotein cholesterol (HDL-c), low density lipoprotein cholesterol (LDL-c), triglyceride, coronary heart disease risk using the Framingham function adapted to Spain and validated in this population and ABI measurement.
Effectiveness: change from baseline on the perceived functional social support | at the study entry and at 12 months.
  The questionnaire Duke-UNC-11 will be used to determine the perceived functional social support.
Effectiveness: change from baseline on anxiety symptoms | at the study entry and at 12 months.
  The General Anxiety Disorder-7 (GAD-7) questionnaire will be used to determine the prevalence and the severity of anxiety symptoms.
Effectiveness: change from baseline on diet quality | at the study entry and at 12 months.
  Diet Quality Index-International (DQI-I) will be used to determine diet quality.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Bolibar-Ribas, MD MSc, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morton K, Beauchamp M, Prothero A, Joyce L, Saunders L, Spencer-Bowdage S, Dancy B, Pedlar C. The effectiveness of motivational interviewing for health behaviour change in primary care settings: a systematic review. Health Psychol Rev. 2015;9(2):205-23. doi: 10.1080/17437199.2014.882006. Epub 2014 Feb 12. PMID 26209209
- [Background] Prestwich A, Webb TL, Conner M. Using theory to develop and test interventions to promote changes in health behaviour: Evidence, issues, and recommendations. Curr Opin Psychol. 2015;5:1-5.
- [Background] Lin JS, O'Connor E, Evans CV, Senger CA, Rowland MG, Groom HC. Behavioral counseling to promote a healthy lifestyle in persons with cardiovascular risk factors: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 Oct 21;161(8):568-78. doi: 10.7326/M14-0130. PMID 25155549
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Powell BJ, McMillen JC, Proctor EK, Carpenter CR, Griffey RT, Bunger AC, Glass JE, York JL. A compilation of strategies for implementing clinical innovations in health and mental health. Med Care Res Rev. 2012 Apr;69(2):123-57. doi: 10.1177/1077558711430690. Epub 2011 Dec 26. PMID 22203646
- [Background] Proctor E, Silmere H, Raghavan R, Hovmand P, Aarons G, Bunger A, Griffey R, Hensley M. Outcomes for implementation research: conceptual distinctions, measurement challenges, and research agenda. Adm Policy Ment Health. 2011 Mar;38(2):65-76. doi: 10.1007/s10488-010-0319-7. PMID 20957426
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N, Wensing M, Fiander M, Eccles MP, Godycki-Cwirko M, van Lieshout J, Jager C. Tailored interventions to address determinants of practice. Cochrane Database Syst Rev. 2015 Apr 29;2015(4):CD005470. doi: 10.1002/14651858.CD005470.pub3. PMID 25923419
- [Background] Ramos R, Baena-Diez JM, Quesada M, Solanas P, Subirana I, Sala J, Alzamora M, Fores R, Masia R, Elosua R, Grau M, Cordon F, Pera G, Rigo F, Marti R, Ponjoan A, Cerezo C, Brugada R, Marrugat J. Derivation and validation of REASON: a risk score identifying candidates to screen for peripheral arterial disease using ankle brachial index. Atherosclerosis. 2011 Feb;214(2):474-9. doi: 10.1016/j.atherosclerosis.2010.11.015. Epub 2010 Nov 19. PMID 21167488
- [Result] Rubio-Valera M, Pons-Vigues M, Martinez-Andres M, Moreno-Peral P, Berenguera A, Fernandez A. Barriers and facilitators for the implementation of primary prevention and health promotion activities in primary care: a synthesis through meta-ethnography. PLoS One. 2014 Feb 28;9(2):e89554. doi: 10.1371/journal.pone.0089554. eCollection 2014. PMID 24586867
- [Result] Zabaleta-del-Olmo E, Bolibar B, Garcia-Ortiz L, Garcia-Campayo J, Llobera J, Bellon JA, Ramos R. Building interventions in primary health care for long-term effectiveness in health promotion and disease prevention. A focus on complex and multi-risk interventions. Prev Med. 2015 Jul;76 Suppl:S1-4. doi: 10.1016/j.ypmed.2015.03.011. Epub 2015 Mar 14. No abstract available. PMID 25778858
- [Result] Fernandez A, Moreno-Peral P, Zabaleta-del-Olmo E, Bellon JA, Aranda-Regules JM, Luciano JV, Serrano-Blanco A, Rubio-Valera M. Is there a case for mental health promotion in the primary care setting? A systematic review. Prev Med. 2015 Jul;76 Suppl:S5-11. doi: 10.1016/j.ypmed.2014.11.019. Epub 2014 Dec 2. PMID 25475684
- [Result] Garcia-Campayo J, del Hoyo YL, Valero MS, Yus MC, Esteban EA, Guedea MP, Botaya RM. Primary prevention of anxiety disorders in primary care: A systematic review. Prev Med. 2015 Jul;76 Suppl:S12-5. doi: 10.1016/j.ypmed.2014.10.015. Epub 2014 Oct 16. PMID 25456801
- [Result] Gili M, Vicens C, Roca M, Andersen P, McMillan D. Interventions for preventing relapse or recurrence of depression in primary health care settings: A systematic review. Prev Med. 2015 Jul;76 Suppl:S16-21. doi: 10.1016/j.ypmed.2014.07.035. Epub 2014 Sep 3. PMID 25192769
- [Result] Bellon JA, Moreno-Peral P, Motrico E, Rodriguez-Morejon A, Fernandez A, Serrano-Blanco A, Zabaleta-del-Olmo E, Conejo-Ceron S. Effectiveness of psychological and/or educational interventions to prevent the onset of episodes of depression: A systematic review of systematic reviews and meta-analyses. Prev Med. 2015 Jul;76 Suppl:S22-32. doi: 10.1016/j.ypmed.2014.11.003. Epub 2014 Nov 20. PMID 25445331
- [Result] Alvarez-Bueno C, Rodriguez-Martin B, Garcia-Ortiz L, Gomez-Marcos MA, Martinez-Vizcaino V. Effectiveness of brief interventions in primary health care settings to decrease alcohol consumption by adult non-dependent drinkers: a systematic review of systematic reviews. Prev Med. 2015 Jul;76 Suppl:S33-8. doi: 10.1016/j.ypmed.2014.12.010. Epub 2014 Dec 13. PMID 25514547
- [Result] Maderuelo-Fernandez JA, Recio-Rodriguez JI, Patino-Alonso MC, Perez-Arechaederra D, Rodriguez-Sanchez E, Gomez-Marcos MA, Garcia-Ortiz L. Effectiveness of interventions applicable to primary health care settings to promote Mediterranean diet or healthy eating adherence in adults: A systematic review. Prev Med. 2015 Jul;76 Suppl:S39-55. doi: 10.1016/j.ypmed.2014.12.011. Epub 2014 Dec 16. PMID 25524613
- [Result] Sanchez A, Bully P, Martinez C, Grandes G. Effectiveness of physical activity promotion interventions in primary care: A review of reviews. Prev Med. 2015 Jul;76 Suppl:S56-67. doi: 10.1016/j.ypmed.2014.09.012. Epub 2014 Sep 26. PMID 25263343
- [Result] Alvarez-Bueno C, Cavero-Redondo I, Martinez-Andres M, Arias-Palencia N, Ramos-Blanes R, Salcedo-Aguilar F. Effectiveness of multifactorial interventions in primary health care settings for primary prevention of cardiovascular disease: A systematic review of systematic reviews. Prev Med. 2015 Jul;76 Suppl:S68-75. doi: 10.1016/j.ypmed.2014.11.028. Epub 2014 Dec 12. PMID 25511466
- [Result] Bully P, Sanchez A, Zabaleta-del-Olmo E, Pombo H, Grandes G. Evidence from interventions based on theoretical models for lifestyle modification (physical activity, diet, alcohol and tobacco use) in primary care settings: A systematic review. Prev Med. 2015 Jul;76 Suppl:S76-93. doi: 10.1016/j.ypmed.2014.12.020. Epub 2015 Jan 5. PMID 25572619
- [Result] March S, Torres E, Ramos M, Ripoll J, Garcia A, Bulilete O, Medina D, Vidal C, Cabeza E, Llull M, Zabaleta-del-Olmo E, Aranda JM, Sastre S, Llobera J. Adult community health-promoting interventions in primary health care: A systematic review. Prev Med. 2015 Jul;76 Suppl:S94-104. doi: 10.1016/j.ypmed.2015.01.016. Epub 2015 Jan 24. PMID 25625691
- [Result] Moreno-Peral P, Conejo-Ceron S, Fernandez A, Berenguera A, Martinez-Andres M, Pons-Vigues M, Motrico E, Rodriguez-Martin B, Bellon JA, Rubio-Valera M. Primary care patients' perspectives of barriers and enablers of primary prevention and health promotion-a meta-ethnographic synthesis. PLoS One. 2015 May 4;10(5):e0125004. doi: 10.1371/journal.pone.0125004. eCollection 2015. PMID 25938509
- [Result] Martin Cantera C, Puigdomenech E, Ballve JL, Arias OL, Clemente L, Casas R, Roig L, Perez-Tortosa S, Diaz-Gete L, Granollers S. Effectiveness of multicomponent interventions in primary healthcare settings to promote continuous smoking cessation in adults: a systematic review. BMJ Open. 2015 Oct 1;5(10):e008807. doi: 10.1136/bmjopen-2015-008807. PMID 26428333
- [Result] Berenguera A, Pons-Vigues M, Moreno-Peral P, March S, Ripoll J, Rubio-Valera M, Pombo-Ramos H, Asensio-Martinez A, Bolanos-Gallardo E, Martinez-Carazo C, Maderuelo-Fernandez JA, Martinez-Andres M, Pujol-Ribera E. Beyond the consultation room: Proposals to approach health promotion in primary care according to health-care users, key community informants and primary care centre workers. Health Expect. 2017 Oct;20(5):896-910. doi: 10.1111/hex.12530. Epub 2017 Jan 24. PMID 28116774
- [Result] Pons-Vigues M, Berenguera A, Coma-Auli N, March S, Pombo H, Masluk B, Pulido-Fuentes M, Rodriguez C, Bellon JA, Pujol-Ribera E. Qualitative evaluation of a complex intervention to implement health promotion activities according to healthcare attendees and health professionals: EIRA study (phase II). BMJ Open. 2019 Mar 23;9(3):e023872. doi: 10.1136/bmjopen-2018-023872. PMID 30904842
- [Result] Pons-Vigues M, Berenguera A, Coma-Auli N, Pombo-Ramos H, March S, Asensio-Martinez A, Moreno-Peral P, Mora-Simon S, Martinez-Andres M, Pujol-Ribera E. Health-care users, key community informants and primary health care workers' views on health, health promotion, health assets and deficits: qualitative study in seven Spanish regions. Int J Equity Health. 2017 Jun 13;16(1):99. doi: 10.1186/s12939-017-0590-2. PMID 28610633
- [Result] Zabaleta-Del-Olmo E, Pombo H, Pons-Vigues M, Casajuana-Closas M, Pujol-Ribera E, Lopez-Jimenez T, Cabezas-Pena C, Martin-Borras C, Serrano-Blanco A, Rubio-Valera M, Llobera J, Leiva A, Vicens C, Vidal C, Campinez M, Martin-Alvarez R, Maderuelo JA, Recio JI, Garcia-Ortiz L, Motrico E, Bellon JA, Moreno-Peral P, Martin-Cantera C, Claveria A, Aldecoa-Landesa S, Magallon-Botaya R, Bolibar B. Complex multiple risk intervention to promote healthy behaviours in people between 45 to 75 years attended in primary health care (EIRA study): study protocol for a hybrid trial. BMC Public Health. 2018 Jul 13;18(1):874. doi: 10.1186/s12889-018-5805-y. PMID 30005705
- [Derived] Sanchez-Recio R, Olivan-Blazquez B, Mendez-Lopez F, Gascon-Santos S, Marti-Lluch R, Zabaleta-Del-Olmo E, Tamayo-Morales O, Maderuelo-Fernandez JA, Casajuana M, Lopez-Jimenez T, Motrico E, Gomez-Gomez I, Sanchez-Perez A, Rodero-Cosano ML, Llobera J, Bellon JA, Moreno-Peral P, Bolibar B, Recio-Rodriguez JI, Ramos R, Claveria A. Self-reported health and depression among EIRA cohort: a moderated mediation model of sex and perceived social support. Front Psychol. 2025 Jun 13;16:1540530. doi: 10.3389/fpsyg.2025.1540530. eCollection 2025. PMID 40584072
- [Derived] Gomez-Gomez I, Motrico E, Moreno-Peral P, Casajuana-Closas M, Lopez-Jimenez T, Zabaleta-Del-Olmo E, Claveria A, LLobera J, Marti-Lluch R, Ramos R, Maderuelo-Fernandez JA, Vicens C, Dominguez-Garcia M, Bartolome-Moreno C, Recio-Rodriguez JI, Bellon JA. A multiple health behaviour change intervention to prevent depression: A randomized controlled trial. Gen Hosp Psychiatry. 2023 May-Jun;82:86-94. doi: 10.1016/j.genhosppsych.2023.02.004. Epub 2023 Feb 22. PMID 37001428
- [Derived] Recio-Rodriguez JI, Garcia-Ortiz L, Garcia-Yu IA, Lugones-Sanchez C, Olmo EZ, Bolibar B, Casajuana-Closas M, Lopez-Jimenez T, Llobera J, Ramos R, Pombo H, Motrico E, Gil-Girbau M, Lopez-Mendez F, Represas-Carrera F, Maderuelo-Fernandez JA. Effectiveness of a multiple health-behaviour-change intervention in increasing adherence to the Mediterranean Diet in adults (EIRA study): a randomized controlled hybrid trial. BMC Public Health. 2022 Nov 19;22(1):2127. doi: 10.1186/s12889-022-14590-y. PMID 36401247
- [Derived] Zabaleta-Del-Olmo E, Casajuana-Closas M, Lopez-Jimenez T, Pombo H, Pons-Vigues M, Pujol-Ribera E, Cabezas-Pena C, Llobera J, Marti-Lluch R, Vicens C, Motrico E, Gomez-Gomez I, Maderuelo-Fernandez JA, Recio-Rodriguez JI, Masluk B, Contreras-Martos S, Jacques-Avino C, Aznar-Lou I, Gil-Girbau M, Claveria A, Magallon-Botaya R, Bellon JA, Ramos R, Sanchez-Perez A, Moreno-Peral P, Leiva A, Gonzalez-Formoso C, Bolibar B. Multiple health behaviour change primary care intervention for smoking cessation, physical activity and healthy diet in adults 45 to 75 years old (EIRA study): a hybrid effectiveness-implementation cluster randomised trial. BMC Public Health. 2021 Dec 4;21(1):2208. doi: 10.1186/s12889-021-11982-4. PMID 34863136
- [Derived] Aznar-Lou I, Zabaleta-Del-Olmo E, Casajuana-Closas M, Sanchez-Vinas A, Parody-Rua E, Bolibar B, Iracheta-Todo M, Bulilete O, Lopez-Jimenez T, Pombo-Ramos H, Martin Miguel MV, Magallon-Botaya R, Maderuelo-Fernandez JA, Motrico E, Bellon J, Marti-Lluch R, Rubio-Valera M, Serrano-Blanco A. Cost-effectiveness analysis of a multiple health behaviour change intervention in people aged between 45 and 75 years: a cluster randomized controlled trial in primary care (EIRA study). Int J Behav Nutr Phys Act. 2021 Jul 2;18(1):88. doi: 10.1186/s12966-021-01144-5. PMID 34215275